CLINICAL TRIAL: NCT00915070
Title: Role of Endothelin-1 in Optic Nerve Head Blood Flow Regulation During Isometric Exercise in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Ass.Prof.Priv.Doz.Dr., Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OPHT-320708
Record Dates: First submitted 2009-06-01; First posted 2009-06-05 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: BQ-123; Optic Nerve Head Blood Flow; Intraocular Pressure; Regional Blood Flow; Ocular Physiology; Optic Disk
MeSH Terms: interventions — cyclo(Trp-Asp-Pro-Val-Leu); Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BQ-123 (Active Comparator)
  Interventions: Drug: BQ-123; Drug: Physiological saline solution; Device: Laser Doppler Flowmetry; Device: Goldmann Applanation Tonometer; Other: squatting
- Physiological saline solution (Placebo Comparator)
  Interventions: Drug: BQ-123; Drug: Physiological saline solution; Device: Laser Doppler Flowmetry; Device: Goldmann Applanation Tonometer; Other: squatting

INTERVENTIONS:
Drug: BQ-123 — 60 mcg/min, infusion period: 60 min
Drug: Physiological saline solution — infusion period 60 minutes
Device: Laser Doppler Flowmetry — blood flow measurements at the temporal neuroretinal rim to assess optic nerve head blood flow
Device: Goldmann Applanation Tonometer — intraocular pressure measurements
Other: squatting — subjects will perform squatting for 6 minutes while blood flow measurements

SUMMARY:
Autoregulation is defined as the ability of a vascular bed to adapt its vascular resistance to changes in perfusion pressure. In the eye, several studies have reported that retinal blood flow is autoregulated over a wide range of ocular perfusion pressures. The investigators could recently show that Endothelin-1 is a key metabolite in the regulation of vascular tone in the eye and plays an important role in the blood flow autoregulation of the choroidal circulation. However, no data is yet available for the optic nerve head. Thus, the present study is designed to test the hypothesis that Endothelin-1 plays also a role in optic nerve head blood flow autoregulation.

Therefore, subjects will perform squatting to increase systemic perfusion pressure during administration of either an endothelin A-receptor blocker (BQ-123) or placebo. Optic nerve head blood flow will be continuously measured during the procedure to investigate optic nerve head autoregulation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years, nonsmokers
* Men and women will be included in equal parts
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal findings in the laboratory testings unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia less than 3 diopters

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except intake of oral contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Optic nerve head pressure-flow relationship | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Univ.Doz, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria